CLINICAL TRIAL: NCT01374074
Title: Racial Disparity in Barrett's Esophagus
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nicholas Shaheen, MD, Professor of Medicine and Epidemiology Director, Center for Esophageal Diseases and Swallowing, University of North Carolina, Chapel Hill
Other Study IDs: 11-0008; U54CA156735 (NIH)
Record Dates: First submitted 2011-06-09; First posted 2011-06-15 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Barrett's Esophagus; Gastroesophageal Reflux Disease (GERD); Intestinal Metaplasia
Keywords: Barrett's Esophagus (BE); Intestinal metaplasia; Gastroesophageal reflux disease (GERD); Racial Disparity
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, plasma, buffy, esophageal biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- White GERD: Participants who self-identify as "not-Hispanic or Latino" and "White" and have been diagnosed by a physician with gastroesophageal reflux disease and do not have Barrett's esophagus.
- African American GERD: Participants who self-identify as "not-Hispanic or Latino" and "African American" and have been diagnosed by a physician with gastroesophageal reflux disease and do no have Barrett's esophagus.
- White BE: Participants who self-identify as "not-Hispanic or Latino" and "White" and have been diagnosed by a physician with Barrett's Esophagus.
- African American BE: Participants who self-identify as "not-Hispanic or Latino" and "African American" and have been diagnosed by a physician with Barrett's Esophagus.

SUMMARY:
The goal of the proposed research is to investigate the molecular mechanisms of racial disparity in Barrett's esophagus (BE), the premalignant lesion of esophageal adenocarcinoma. Specifically, the investigators hypothesize that environmental factors, genetic factors, and potentially gene environment interactions play crucial roles in the observed racial disparity in developing Barrett's esophagus.

Patients are recruited through UNC hospitals prior to scheduled esophagogastroduodenoscopy (EGD). Participants complete a questionnaire, have body measurements obtained, and have blood, biopsies, and gastric aspirate collected. Participants also complete a 24 hour pH impedance test.

DETAILED DESCRIPTION:
The goal of the proposed research is to investigate the molecular mechanisms of racial disparity in Barrett's esophagus, the premalignant lesion of esophageal adenocarcinoma. Specifically, the investigators hypothesize that environmental factors, genetic factors, and potentially gene environment interactions play crucial roles in the observed racial disparity in developing Barrett's esophagus.

Participants: Patients aged 18-80 presenting at the Gastrointestinal (Gl) Endoscopy Clinic at UNC-Chapel Hill for elective upper endoscopy with a primary or secondary indication of reflux symptoms.

Procedures (methods): Endoscopic biopsy, pH impedance and sampling of gastric secretions will be performed according to our standard protocol. A series of questionnaires assessing demographics, environmental exposure (e.g., smoking, drinking), markers of socioeconomic status (SES), body measurement, previous health history, and gastroesophageal reflux disease (GERD) symptomatology will be administered to our subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80
* Self-identify is "not Hispanic or Latino" and either "African American" or "White."
* Cases will be eligible for inclusion if they have endoscopically evident Barrett's Esophagus (BE) of any length. BE will be defined as: 1) Any upward displacement of the squamocolumnar junction noted on endoscopy such that the interface of squamous and columnar mucosa is no longer at the interface of the most distal tubular esophagus and the proximal gastric folds. The characteristic pale pink coloration of the squamous epithelium in these areas will be replaced by the darker salmon color commonly seen in BE. 2) Histologic interpretation of biopsies consistent with intestinal columnar metaplasia containing goblet cells, which are positively stained by Alcian blue staining as barrel-shaped cells.
* Controls will be eligible for inclusion if they have classic symptoms of gastroesophageal reflux disease (GERD), but no endoscopic or histological evidence of BE. Both erosive and non-erosive GERD will be eligible. Because we expect GERD to outnumber BE and patients with GERD may be slightly less willing to participate in the study than patients with BE (based on recruitment for the studies noted above), we plan to randomly sample one fourth of eligible controls. If approximately 20% fewer GERD than BE participate, a final study population with an approximately 1:2 BE to GERD ratio will be achieved. Oversampling of patients with GERD will improve study power.

Exclusion Criteria:

* Patients who are unable to read or comprehend the informed consent or written questionnaires;
* Patients who are status post partial or complete esophageal resection;
* Patients with prevalent BE who have undergone endoscopic ablation;
* Patients found to have high-grade dysplasia or esophageal cancer on the index endoscopy;
* Patients with surgical anti-reflux procedures;
* Patients of races other than Caucasian and African Americans;
* Pregnant women.
* Patients with a bleeding diathesis or other contraindication of endoscopic biopsy.
* Current use of warfarin, heparin, and/or low molecular weight heparin (requires discontinuation of medication 5 days prior to and 7 days after EGD).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source of the study population will be patients aged 18-80 presenting at the gastrointestinal (Gl) Endoscopy Clinic at UNC-Chapel Hill for elective upper endoscopy with a primary or secondary indication of reflux symptoms. Any patient undergoing endoscopy with classic reflux symptoms is eligible to participate in the study. These symptoms include a substernal chest burning or warmth, a "waterbrash" sensation, regurgitation, or any chest pain worst when supine or after meals.
  Race will be self-identified race or ethnicity (SIRE) from a researcher-provided list. According to the NIH Policy on Reporting Race and Ethnicity Data published in August 8, 2001 (NOT-OD-01-053), we will "use two separate questions with ethnicity information collected first followed by the option to select more than one racial designation." Patients in this study should be "Not Hispanic or Latino", and either "African American" or "White".
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2011-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To examine the association between BE and environmental factors | Enrollment (day 1)
  Odds ratios (ORs) and 95% confidence intervals (CI) will be used to estimate the association between gastroesophageal reflux disease (GERD) and Barrett's esophagus (BE) among Caucasian Americans and African Americans, separately, in relation to patterns of the exposures of interest (tobacco use, alcohol consumption, fruit and vegetable intake and other dietary measures, no NSAID use, and various measures of SES), with adjustments made for the frequency matching factors, age at reference (date of diagnosis for cases and date of identification for controls) and sex.

SECONDARY OUTCOMES:
To investigate the association between BE and genetic and epigenetic status of Cdx1/Cdx2 | Enrollment (day 1)
  The promoter regions of Cdxl and Cdx2 genes will be examined for single nucleotide polymorphisms (SNPs). Pyrosequencing will be used to quantitatively determine the methylation status of Cdxl and Cdx2 promoters in esophageal biopsy tissues. For the single functional genotype analyses, conventional unconditional logistic regression will be used and ORs will be estimated for "at-risk" homozygotes and heterozygotes relative to "wild-type" homozygotes by creating indicator variables for each genotype.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Xiaoxin Chen, MD, PhD, Principal Investigator — North Carolina Central University
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States